CLINICAL TRIAL: NCT00635141
Title: The Effect of Inhaled Hypertonic Saline (7%) Versus Normal Saline (0.9%) on the Lung Clearance Index in Patients With Cystic Fibrosis
Brief Title: The Effect of Hypertonic Saline on the Lung Clearance Index in Patients With Cystic Fibrosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Canadian Cystic Fibrosis Foundation (Other)
Responsible Party: Principal Investigator, Felix Ratjen, Division Head, Respiratory Medicine, The Hospital for Sick Children
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 1000011193
Record Dates: First submitted 2008-03-04; First posted 2008-03-13 (Estimated); Last update posted 2013-09-02 (Estimated); Status verified 2013-08

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis; Lung Clearance Index; Hypertonic Saline; Pediatrics
MeSH Terms: conditions — Cystic Fibrosis | interventions — Saline Solution, Hypertonic; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: hypertonic saline (7 %) and isotonic saline (0.9%)
- 2 (Experimental)
  Interventions: Drug: hypertonic saline (7 %) and isotonic saline (0.9%)

INTERVENTIONS:
Drug: hypertonic saline (7 %) and isotonic saline (0.9%) — Patients in study arm 1 will receive hypertonic saline (7 %) during the first phase of the study and will crossover to placebo (0.9% isotonic saline) during the second phase. Both drugs will be administered via PARI LC® Star reusable nebulizer.
  Arms: 1
Drug: hypertonic saline (7 %) and isotonic saline (0.9%) — Patients in study arm 2 will receive placebo (0.9% isotonic saline) during the first phase of the study and will crossover to hypertonic saline (7 %) during the second phase. Both drugs will be administered via PARI LC® Star reusable nebulizer.
  Arms: 2

SUMMARY:
This study is examining the effect of hypertonic saline compared to placebo on the Lung Clearance Index in Cystic Fibrosis patients.

DETAILED DESCRIPTION:
The life expectancy of patients with Cystic Fibrosis (CF) has greatly increased over time due to improved clinical care. While this is certainly beneficial to CF patients, the overall stability in lung function has made it more difficult to assess the effect of therapeutic interventions. Currently, FEV1 (forced expiratory volume in 1 second) remains the primary outcome measure for most clinical trials, but many CF patients have normal pulmonary function and the annual rate of decline is now less than 2% in large specialized centres. Therefore, additional parameters are needed that are more sensitive parameters to define abnormalities in CF patients and be used in therapeutic trials.

One such promising parameter is the Lung Clearance Index (LCI). The LCI is a test to quantify ventilation inhomogeneity by assessing the washout of an inhaled inert gas. Abnormalities in gas clearance from the lung are largely due to retention of inhaled gases due to mucous obstruction in the lower airways.

Interventions that improve mucus accumulation are expected to improve the LCI. Hypertonic saline has been shown to increase airway surface liquid (ASL), mucociliary clearance and pulmonary function. Therefore, this study will examine the effect of hypertonic saline compared to placebo on the Lung Clearance Index in Cystic Fibrosis patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CF as defined by two or more clinical features of CF and a documented sweat chloride > 60 mEq/L by quantitative pilocarpine iontophoresis test or a genotype showing two well characterized disease causing mutations
* Informed consent and verbal assent (as appropriate) provided by the subject's parent or legal guardian and the subject
* 6-18 years of age at enrolment and able to perform reproducible spirometry
* Clinically stable at enrolment
* FEV1 % predicted ≥ 80 % as calculated by the Wang reference equations
* Ability to comply with medication use, study visits and study procedures

Exclusion Criteria:

* Respiratory culture positive for NTM or B. cepacia complex within past year or screening
* Use of intravenous antibiotics or oral quinolones within 14 days of screening
* Investigational drug use within 30 days of screening
* Physical findings at screening that would compromise the safety of the participant or the quality of the study data

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2008-03; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Change in LCI from baseline to end of treatment in hypertonic saline treated patients versus patients receiving placebo (isotonic saline) | Duration of patient's involvement in study

SECONDARY OUTCOMES:
Change in FEV1 % predicted | Duration of patient's involvement in study
Change in FVC (forced vital capacity) % predicted | Duration of patient's involvement in study
Change in FEF25-75% (forced expiratory flow between 25 and 75 % of vital capacity) predicted | Duration of patient's involvement in study

CONTACTS AND LOCATIONS:
Overall Officials: Felix Ratjen, MD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

REFERENCES:
- [Result] Amin R, Subbarao P, Jabar A, Balkovec S, Jensen R, Kerrigan S, Gustafsson P, Ratjen F. Hypertonic saline improves the LCI in paediatric patients with CF with normal lung function. Thorax. 2010 May;65(5):379-83. doi: 10.1136/thx.2009.125831. PMID 20435858
- [Derived] Wark P, McDonald VM, Smith S. Nebulised hypertonic saline for cystic fibrosis. Cochrane Database Syst Rev. 2023 Jun 14;6(6):CD001506. doi: 10.1002/14651858.CD001506.pub5. PMID 37319354